CLINICAL TRIAL: NCT05461339
Title: A Phase III, Randomized, Multicenter, Doubled-blind Clinical Trial Comparing the Efficacy and Safety of TAB014 and Lucentis in Neovascular Age-related Macular Degeneration (nAMD) Patients
Brief Title: TAB014 Compared to Lucentis® in Patients with Neovascular Age-related Macular Degeneration
Acronym: nAMD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioDlink Biopharm Co., Ltd. (Industry)
Collaborators: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOT-CR-TAB014-III-01
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators responsible for patient care, vision examiner (including BCVA assessors), research nurses, independent central reading center staff, and the sponsor are blinded. Unmasked pharmacist, unmasked nurse, unmasked treatment administration physician and unmasked research associates will take part in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAB014 (Experimental): intravitreal injection at 1.25mg once every 4 week
  Interventions: Drug: TAB014 Monoclonal Antibody Injection
- Ranibizumb (Active Comparator): intravitreal injection at 0.5mg once every 4 week
  Interventions: Drug: Ranibizumab Injection [Lucentis]

INTERVENTIONS:
Drug: TAB014 Monoclonal Antibody Injection — intravitreal injection at 1.25mg once every 4 weeks
  Other Names: TAB014
  Arms: TAB014
Drug: Ranibizumab Injection [Lucentis] — intravitreal injection at 0.5mg once every 4 weeks
  Other Names: Lucentis
  Arms: Ranibizumb

SUMMARY:
This study is a randomized, multi-center, double blind, Lucentis controlled non-inferiority study in neovascular age-related macular degeneration patients. The objective of this study is to compare the efficacy and safety of TAB014 and ranibizumab (Lucentis).

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the efficacy of TAB014 compared to Lucentis in neovascular age-related macular degeneration patients

Secondary Objectives:

1. To evaluate the safety of TAB014 compared to Lucentis in neovascular age-related macular degeneration patients.
2. To evaluate the immunogenicity of TAB014 in neovascular age-related macular degeneration patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be > 50 years old, male or female;
2. Confirmed active subfoveal or juxtafoveal choroidal neovascularization (CNV) secondary to nAMD in the study eye;
3. BCVA letter score between 15 and 73 (inclusive) by the ETDRS chart during the screening period ;
4. Confirmed by independent central reading center:

   1. Total lesion area ≤ 12 optic disc areas in the study eye,
   2. Fibrotic, scarring or atrophy < 50% of total lesion area, without involving the fovea,
   3. Retinal hemorrhage involving the foveal or intraretinal hemorrhage < 4 optic disc area,
5. Able to understand and personally sign informed consent form.

Exclusion Criteria:

1. Ophthalmic Treatment history:

   1. Intravitreal injection of an anti-VEGF drug (ranibizumab, bevacizumab, aflibercept or conbercept, etc.) in any eye within 90 days prior to randomization;
   2. Prior vitrectomy, panretinal photocoagulation, laser treatment of the foveal area or ocular treatment/surgery for nAMD in the study eye; or history of corneal transplantation or corneal dystrophy, treatment with verteporfin, external radiation therapy of the head or the eye, transpupillary hyperthermia;
   3. Prior intra-ocular (including cataract) surgery in the study eye within 90 days before randomization, or surgery to the exterior eye within 28 days before randomization;
   4. Intravitreal therapy in the study eye (e.g. steroids or device implants) within 180 days before randomization;
   5. PDT (Photodynamic Therapy) in the non-study eye within 30 days before screening;
   6. Central serous chorioretinopathy (CSC) in the study eye;
2. The non-study eye confirmed to have a BCVA on ETDRS chart of < 18 letters during screening;
3. Myopia more than -8.0 diopters of refractive error in study eye; For patients who have undergone refractive surgery or cataract surgery, refraction must not have been greater than -8.0 diopters prior to surgery;
4. Absence of the crystalline lens (unless there has been artificial lens replacement), or presence of posterior lens capsule rupture, or YAG laser posterior capsulotomy received 30 days before randomization or expect to receive during the study period in study eye;
5. Ocular disorders in the study eye as determined by the investigator at the present time: (a) effects on the central vision, or (b) increasing safety risk for the subject, or (c) affecting efficacy, safety evaluation or sampling, or (d) having ocular diseases requiring surgical or medical intervention
6. In the study eye, (a) presence of uncontrolled glaucoma at randomization, or (b) prior glaucoma surgery, or (c) advanced glaucoma or optic neuropathy, affecting or endangering the central visual field;
7. Active intraocular, extraocular, or periocular inflammation or infection in either eye at randomization;
8. History of idiopathic or autoimmune-associated uveitis in either;
9. Active Hepatitis B, C or syphillis; HIV antibody positive; presence of any immune deficient, and/or immune suppressed illnesses;
10. Poorly controlled hypertension after receiving the best possible therapy;
11. Diabetic patients with HbA1c >10%;
12. Any unmanageable clinical illness; Severe liver and kidney abnormalities；dysfunction of blood coagulation; cardiovascular events within 180 days before randomization and determined by investigator can affect subject safety evaluation or increase subject risk;
13. Prior significant allergic reactions to biological products, or known allergic reactions to bevacizumab, ranibizumab, or study related medication (including fluorescein or indocyanin green), pupillary dilating agents, anaesthetic agents, or anti-infective agents;
14. Anti-VEGF therapy within 90 days prior to randomization; subjects are allowed to take any dietary supplements, vitamins or minerals;
15. Continuous systemic use ≥ 30days of corticosteroids within 90 days before randomization, or systemic use of corticosteroids within 5 days before randomization;
16. Necessity to continue use of prohibited agents (drugs known to be toxic to the lens, retina, or optic nerve, including deoxyamine, chloroquine/hydroxychloroquine (braquinib), tamoxifen, phenothiazines, and ethambutol);
17. Participation in a study trial involving any drug or device therapy (other than vitamins and minerals) within 90 days prior to randomization; And the use of any other experimental drugs or experimental interventions other than those of this study (e.g. isostoluent blood thinning, intravitreal tissue plasminogen activators) is prohibited during the study period;
18. Pregnant or lactating women, or those with plans for pregnancy during or within 6 months of study termination (including male subjects). Premenopausal woman testing positive for pregnancy during screening or is reluctant to use reliable contraceptive methods during the study periods;
19. Other conditions that are considered not acceptable to be enrolled in the study by the investigator.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in BCVA of the study eye from TAB014 and ranibizumab treatment groups. | At week 52
  Best-corrected visual acuity (BCVA) letter score as measured by the ETDRS chart

SECONDARY OUTCOMES:
Evaluate the change in BCVA of the study eye | At week 12, 24 and 36
  Best-corrected visual acuity (BCVA) letter score as measured by the ETDRS chart
Evaluate the proportion of subjects with an increase in BCVA of >5, >10, and >15 in the study eye | At week 12, 24 and 52
  Best-corrected visual acuity (BCVA) letter score as measured by the ETDRS chart
Evaluate the proportion of subjects with a BCVA loss of <5, <10, < 15 letters in the study eye | At week 12, 24 and 52
  Best-corrected visual acuity (BCVA) letter score as measured by the ETDRS chart
Change in central subfield thickness（CST) in the study eye | At week 12, 24, 36 and 52
  CST measured by SD-OCT as assessed by independent central reading center
Change in Choroidal Neovascularization (CNV) area of study eye | At week 12, 24 and 52
  CNV as assessed by independent central reading center

OTHER OUTCOMES:
Safety Evaluation | Baseline and every month up to week 52
  Ocular and non-ocular adverse events, serious adverse events (SAEs), adverse events of special interest (AESI), etc. will be graded according to the Ophthalmic Adverse Event Grading Scale and NIA Guidelines for Adverse Events and Serious Adverse Events (September 2018 Edition).
Immunogenicity Evaluation | At week 12, 24 and 52
  Detection of anti-drug antibody and/or neutralizing antibodies will be examined in approximately 80 patients with monocular nAMD and no prior anti-VEGF therapy in the non-study eye for detection of immunogenicity evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (56):
- China (56):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Aier Intech Eye Hospital, Beijing, Beijing Municipality
  - Peking University People'S Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Cmu, Beijing, Beijing Municipality
  - The First Hospital of Jilin University, Jilin, Changchun
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong
  - Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong, Shantou, Guangdong
  - Shenzhen Aier Eye Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Eye Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Kaifeng Central Hopital, Kaifeng, Henan
  - Henan Eye Hospital& Henan Eye Institute, Zhengzhou, Henan
  - Zhengzhou Second Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital (Affiliated Hospital of Hubei University of Medicine), Shiyan, Hubei
  - Tongji Hospital® Tongji Medical Collehe of Hust, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Central theater General Hospital, Wuhan, Hubei
  - Wuhan Puren Hospital, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Aier Eye Hospital(Changsha), Changsha, Hunan
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Dalian No.3 People'S Hospital, Dalian, Liaoning
  - The Fourth People's Hospital of Shenyang, Shenyang, Liaoning
  - Shenyang He Eye Hospital, Shenyang, Liaoning
  - Weifang Eye Hospital Co., Ltd., Weifang, Shandong
  - Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital(Tenth People's Hospital of Tongji Unversity), Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Changzhi People'S Hospital, Changzhi, Shanxi
  - The First People's Hospital of Jinzhong(Jinzhong Hospital Affiliated to Shanxi Medical University), Jinzhong, Shanxi
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Xi'an No.1 Hospital, Xi’an, Shanxi
  - Xi'An Fourth Hospital, Xi’an, Shanxi
  - Chengdu Aier Eye Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Ineye Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU), Hangzhou, Zhejiang
  - Zhejiang Provincial People'S Hospital, Hangzhou, Zhejiang
  - Eye Hospital, WMU, Wenzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No